CLINICAL TRIAL: NCT01231789
Title: The Neuroprotection of Remote Ischemic Preconditioning on Cardiac Surgery in Multicenter
Brief Title: The Neuroprotection of Remote Ischemic Preconditioning (RIPC) on Cardiac Surgery in Multicenter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RIPC-Cardiac-Neuroprotection
Record Dates: First submitted 2010-09-15; First posted 2010-11-01 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2009-06

CONDITIONS: Cardiac Surgery Patients
Keywords: cardiac surgery; RIPC; brain injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sham RIPC (Sham Comparator): Patients had a deflated cuff placed on the right upper arm for 30 min.
  Interventions: Procedure: sham RIPC
- RIPC treatment (Experimental): RIPC consisted of three 5-min cycles of right upper arm ischemia, which was induced by an automated cuff-inflator placed on the right upper arm and inflated to 200 mmHg, with an intervening 5 min of reperfusion during which the cuff was deflated
  Interventions: Procedure: RIPC

INTERVENTIONS:
Procedure: RIPC — RIPC consisted of three 5-min cycles of right upper arm ischemia, which was induced by an automated cuff-inflator placed on the right upper arm and inflated to 200 mmHg, with an intervening 5 min of reperfusion during which the cuff was deflated
  Other Names: remote ischemic preconditioning
  Arms: RIPC treatment
Procedure: sham RIPC — Patients had a deflated cuff placed on the right upper arm for 30 min without any inflation procedure.
  Other Names: sham remote ischemic preconditioning
  Arms: sham RIPC

SUMMARY:
The current study is designed to clarify the neuroprotective effect of remote ischemic preconditioning on the patients underwent open-heart cardiac surgery.

DETAILED DESCRIPTION:
BACKGROUND: Brain ischemia and injury are commonly contributed to perioperative morbidity and mortality after cardiac surgery. Remote ischemic preconditioning (RIPC) is a phenomenon whereby brief periods of ischemia followed by reperfusion in one organ provide systemic protection from prolonged ischemia. To investigate whether remote preconditioning protects the brain injury in patients undergoing elective cardiac surgery, a randomized trial will be performed in current study.

DESIGNING 150 patients will be randomize assigned to cardiac surgery with RIPC or without RIPC (control). Remote ischemic preconditioning consist of three 5-min cycles of right upper limb ischaemia, induced by an automated cuff-inflator placed on the upper arm and inflated to 200 mm Hg, with an intervening 5 min of reperfusion during which the cuff is deflated. Cerebral injury was assessed by S-100b, NSE, and neurological function scores in different time points.

EXPECTED RESULTS RIPC will reduce the incidence of cerebral injury in cardiac surgery.

CONCLUSIONS:

In patients undergoing elective cardiac surgery, RIPC reduces the incidence of postoperative cerebral injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acquired heart valve diseases scheduled for valve replacement or CABG

Exclusion Criteria:

* Were unable to give informed consent
* Patients who presented with other systemic diseases such as hepatic,renal, and pulmonary diseases, or have had a heart operation before, were excluded.
* Additionally, patients taking antidiabetic sulfonylurea or glibenclamide were excluded because these agents have been shown to abrogate the cardioprotection elicited by ischemic preconditioning.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
the neurological injury markers, including serum level of S-100B and NSE | before surgery, 6h, 24h, 48h, and 72h after bypass
  the biomarkers of brain injury

SECONDARY OUTCOMES:
mini-mental state examination scale | 6 months after surgery
  the neurological function

CONTACTS AND LOCATIONS:
Overall Officials: Hailong Dong, MD,PhD, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Zhu S, Zheng Z, Lv W, Ouyang P, Han J, Zhang J, Dong H, Lei C. Neuroprotective effect of remote ischemic preconditioning in patients undergoing cardiac surgery: A randomized controlled trial. Front Cardiovasc Med. 2022 Sep 6;9:952033. doi: 10.3389/fcvm.2022.952033. eCollection 2022. PMID 36148077